CLINICAL TRIAL: NCT05455229
Title: Elucidating How Physical Activity and Sleep Relate to Optimal Cognitive Ageing: the PASOCA- Study
Brief Title: Elucidating How Physical Activity and Sleep Relate to Optimal Cognitive Ageing
Acronym: PASOCA
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: University Ghent (Other); Research Foundation Flanders (Other)
Responsible Party: Principal Investigator, Pieter-Jan Marent, Principal Investigator, KU Leuven
Other Study IDs: PASOCA_2021
Record Dates: First submitted 2021-11-08; First posted 2022-07-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Cognitive Aging
Keywords: Physical activity; Sedentary behaviour; Sleep; Cognition; Ageing; Longitudinal; Observational; Accelerometry
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Increased longevity is one of the greatest success stories in public health. However, ageing is accompanied by cognitive decline which affects people's daily functioning and, if it develops to dementia, their ability to live independently. By 2050, the number of people who develop dementia will triple to 152 million. The aim of this project is to precisely examine how physical activity (PA) and sleep, both modifiable lifestyle factors, are related to cognitive function and which role they can play in optimal cognitive ageing. To do so, a longitudinal study will be conducted, with objective measures of PA, sleep and cognition in midlife and older adults. This project will meet the current need for longitudinal studies with objective PA and sleep data, as well as provide, for the first time, in-depth information on associations of type of PA (aerobic vs muscle strengthening), characteristics of sleep (quality vs quantity) with specific cognitive domains (executive function and memory). Furthermore, although PA and sleep are related, the behavioural dynamics of combinations of PA and sleep on cognition has never been studied before. To fill this gap, these relationships will be examined with an innovative statistical approach, looking at data across a 24-hour period. The resulting deeper understanding of the precise relationship between PA, sleep and cognitive function will contribute to the development of preventive interventions for maintaining cognitive health at older age.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling, healthy adults aged 55 and above

Exclusion Criteria:

1. has a neurodegenerative disease such as Parkinson's, Alzheimer's, MS…; or
2. has a psychiatric illness such as bipolar disorder, OCD…; or
3. has had a serious brain injury in the past year or before that is still affecting them; or
4. has had a brain haemorrhage; or
5. is currently experiencing a depressive episode; or
6. has a history of addiction or excessive alcohol abuse; or
7. uses a sleeping device (for sleep apnoea); or
8. has chronic insomnia (diagnosed insomnia); or
9. is severely limited in performing daily activities (up and down stairs, walk ...)
10. has a first-degree dementia within the family
11. scores a 23 or lower on the Montreal Cognitive Assessment

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community dwelling, healthy adults aged 55 and above living in Belgium.
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Cognitive function (baseline) - objective: executive function and memory will be tested with Cambridge Neuropsychological Test Automated Battery (CANTAB) | baseline
  Executive functions and memory will be the main outcome measure for cognitive function. Executive control (planning, shifting, inhibiting, attention) and memory (visuospatial, episodic, verbal) functions will be measured objectively using an iPad with the validated CANTAB software (cambridgecognition.com). Specific tasks in the test battery:
  * Practice: MOT (Motor Screening Task)
  * Memory: PAL (Paired Associates Learning), DMS (Delayed Matching to Sample), VRM (Verbal Recognition Memory)
  * Executive control: MTT Multitasking Test, OTS (One Touch Stockings of Cambridge), SWM (Spatial Working Memory)
Change in cognitive function (follow up 1) - objective: executive function and memory will be tested with Cambridge Neuropsychological Test Automated Battery (CANTAB) | 1 year after baseline
  Executive functions and memory will be the main outcome measure for cognitive function. Executive control (planning, shifting, inhibiting, attention) and memory (visuospatial, episodic, verbal) functions will be measured objectively using an iPad with the validated CANTAB software (cambridgecognition.com). Specific tasks in the test battery:
  * Practice: MOT (Motor Screening Task)
  * Memory: PAL (Paired Associates Learning), DMS (Delayed Matching to Sample), VRM (Verbal Recognition Memory)
  * Executive control: MTT Multitasking Test, OTS (One Touch Stockings of Cambridge), SWM (Spatial Working Memory)
Change in cognitive function (follow up 2) - objective: executive function and memory will be tested with Cambridge Neuropsychological Test Automated Battery (CANTAB) | 1 year after follow up 1; 2 years after baseline
  Executive functions and memory will be the main outcome measure for cognitive function. Executive control (planning, shifting, inhibiting, attention) and memory (visuospatial, episodic, verbal) functions will be measured objectively using an iPad with the validated CANTAB software (cambridgecognition.com). Specific tasks in the test battery:
  * Practice: MOT (Motor Screening Task)
  * Memory: PAL (Paired Associates Learning), DMS (Delayed Matching to Sample), VRM (Verbal Recognition Memory)
  * Executive control: MTT Multitasking Test, OTS (One Touch Stockings of Cambridge), SWM (Spatial Working Memory)
Cognitive function (baseline) - subjective: Cognitive Failure Questionnaire | baseline
  25-items will be used to measure subjective cognitive decline by assessing self-reported frequency of failures in several cognitive domains.
Change in cognitive function (follow up 1) - subjective: Cognitive Failure Questionnaire | 1 year after baseline
  25-items will be used to measure subjective cognitive decline by assessing self-reported frequency of failures in several cognitive domains.
Change in cognitive function (follow up 2) - subjective: Cognitive Failure Questionnaire | 1 year after follow up 1; 2 years after baseline
  25-items will be used to measure subjective cognitive decline by assessing self-reported frequency of failures in several cognitive domains.
Sleep (baseline) - objective: accelerometery - characteristic 1: total sleep time | baseline
  Specifically ActiGraph's wGT3X-BT Activity Monitor (ActiGraph, Pensacola, FL). Placement at the wrist results in the increased wear time and accuracy of sleep measurement. Total sleep time is measured in minutes.
Sleep (baseline) - objective: accelerometery - characteristic 2: wake after sleep onset | baseline
  Specifically ActiGraph's wGT3X-BT Activity Monitor (ActiGraph, Pensacola, FL). Placement at the wrist results in the increased wear time and accuracy of sleep measurement. Wake after sleep onset is measured in minutes.
Sleep (baseline) - objective: accelerometery - characteristic 3: sleep efficiency | baseline
  Specifically ActiGraph's wGT3X-BT Activity Monitor (ActiGraph, Pensacola, FL). Placement at the wrist results in the increased wear time and accuracy of sleep measurement. Sleep efficiency is displayed in percentage.
Sleep (baseline) - objective: accelerometery - characteristic 4: sleep latency | baseline
  Specifically ActiGraph's wGT3X-BT Activity Monitor (ActiGraph, Pensacola, FL). Placement at the wrist results in the increased wear time and accuracy of sleep measurement. Sleep latency is measured in minutes.
Change in sleep (follow up 1) - objective: accelerometery - characteristic 1: total sleep time | 1 year after baseline
  Specifically ActiGraph's wGT3X-BT Activity Monitor (ActiGraph, Pensacola, FL). Placement at the wrist results in the increased wear time and accuracy of sleep measurement. Total sleep time is measured in minutes.
Change in sleep (follow up 1) - objective: accelerometery - characteristic 2: wake after sleep onset | 1 year after baseline
  Specifically ActiGraph's wGT3X-BT Activity Monitor (ActiGraph, Pensacola, FL). Placement at the wrist results in the increased wear time and accuracy of sleep measurement. Wake after sleep onset is measured in minutes.
Change in sleep (follow up 1) - objective: accelerometery - characteristic 3: sleep efficiency | 1 year after baseline
  Specifically ActiGraph's wGT3X-BT Activity Monitor (ActiGraph, Pensacola, FL). Placement at the wrist results in the increased wear time and accuracy of sleep measurement. Sleep efficiency is displayed in percentage.
Change in sleep (follow up 1) - objective: accelerometery - characteristic 4: sleep latency | 1 year after baseline
  Specifically ActiGraph's wGT3X-BT Activity Monitor (ActiGraph, Pensacola, FL). Placement at the wrist results in the increased wear time and accuracy of sleep measurement. Sleep latency is measured in minutes.
Change in sleep (follow up 2) - objective: accelerometery - characteristic 1: total sleep time | 1 year after follow up 1; 2 years after baseline
  Specifically ActiGraph's wGT3X-BT Activity Monitor (ActiGraph, Pensacola, FL). Placement at the wrist results in the increased wear time and accuracy of sleep measurement. Total sleep time is measured in minutes.
Change in sleep (follow up 2) - objective: accelerometery - characteristic 2: wake after | 1 year after follow up 1; 2 years after baseline
  Specifically ActiGraph's wGT3X-BT Activity Monitor (ActiGraph, Pensacola, FL). Placement at the wrist results in the increased wear time and accuracy of sleep measurement. Wake after sleep onset is measured in minutes.
Change in sleep (follow up 2) - objective: accelerometery - characteristic 3: sleep efficiency | 1 year after follow up 1; 2 years after baseline
  Specifically ActiGraph's wGT3X-BT Activity Monitor (ActiGraph, Pensacola, FL). Placement at the wrist results in the increased wear time and accuracy of sleep measurement. Sleep efficiency is displayed in percentage.
Change in sleep (follow up 2) - objective: accelerometery - characteristic 4: sleep latency | 1 year after follow up 1; 2 years after baseline
  Specifically ActiGraph's wGT3X-BT Activity Monitor (ActiGraph, Pensacola, FL). Placement at the wrist results in the increased wear time and accuracy of sleep measurement. Sleep latency is measured in minutes.
Sleep (baseline) - subjective: Pittsburgh Sleep Quality Index (PSQI) | Baseline
  The PSQI is a reliable and validated self-report questionnaire that examines the quality of sleep in the past month. It contains of 19 self-rated questions and 5 questions rated by the bed partner or roommate (if available), covering seven sleep areas: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
Change in sleep (follow up 1) - subjective: Pittsburgh Sleep Quality Index (PSQI) | 1 year after baseline
  The PSQI is a reliable and validated self-report questionnaire that examines the quality of sleep in the past month. It contains of 19 self-rated questions and 5 questions rated by the bed partner or roommate (if available), covering seven sleep areas: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
Change in sleep (follow up 2) - subjective: Pittsburgh Sleep Quality Index (PSQI) | 1 year after follow up 1; 2 years after baseline
  The PSQI is a reliable and validated self-report questionnaire that examines the quality of sleep in the past month. It contains of 19 self-rated questions and 5 questions rated by the bed partner or roommate (if available), covering seven sleep areas: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
Physical activity & Sedentary behaviour (baseline) - objective: accelerometery 1 | baseline
  ActiGraph's wGT3X-BT Activity Monitor (ActiGraph, Pensacola, FL) will be used. It measures time spent in different intensities of physical activity as well as sedentary behaviour and sleep. Participants will be asked to wear the accelerometer continuously during seven consecutive days, day and night, at their non-dominant wrist. In addition to wearing the accelerometer, participants will be asked to fill in a daily succinct diary with: (1) bed times, nap times; (2) non-wear times during the day; and (3) specification of most seated activity. These data will be used to complete and to explain gaps in the data set later on in the software programme. The following PA outcomes will be extracted from the ActiGraph data: average time spent per day in sedentary behaviour, light PA and moderate to vigorous PA.
Physical activity & Sedentary behaviour (baseline) - objective: accelerometery 2 | baseline
  A second accelerometer will be placed on the right thigh, namely the activPAL (PAL Technologies Ltd, Glasgow, UK). This device measures postures due to its static acceleration and inclination features. It can quantify postural allocation - which is not possible with the ActiGraph - and is completely waterproof. The following additional PA outcomes will be extracted: time spent sitting/lying, standing, and walking.
Change in Physical activity & Sedentary behaviour (follow up 1) - objective: accelerometery 1 | 1 year after baseline
  ActiGraph's wGT3X-BT Activity Monitor (ActiGraph, Pensacola, FL) will be used. It measures time spent in different intensities of physical activity as well as sedentary behaviour and sleep. Participants will be asked to wear the accelerometer continuously during seven consecutive days, day and night, at their non-dominant wrist. In addition to wearing the accelerometer, participants will be asked to fill in a daily succinct diary with: (1) bed times, nap times; (2) non-wear times during the day; and (3) specification of most seated activity. These data will be used to complete and to explain gaps in the data set later on in the software programme. The following PA outcomes will be extracted from the ActiGraph data: average time spent per day in sedentary behaviour, light PA and moderate to vigorous PA.
Change in Physical activity & Sedentary behaviour (follow up 1) - objective: accelerometery 2 | 1 year after baseline
  A second accelerometer will be placed on the right thigh, namely the activPAL (PAL Technologies Ltd, Glasgow, UK). This device measures postures due to its static acceleration and inclination features. It can quantify postural allocation - which is not possible with the ActiGraph - and is completely waterproof. The following additional PA outcomes will be extracted: time spent sitting/lying, standing, and walking.
Change in Physical activity & Sedentary behaviour (follow up 2) - objective: accelerometery 1 | 1 year after follow up 1; 2 years after baseline
  ActiGraph's wGT3X-BT Activity Monitor (ActiGraph, Pensacola, FL) will be used. It measures time spent in different intensities of physical activity as well as sedentary behaviour and sleep. Participants will be asked to wear the accelerometer continuously during seven consecutive days, day and night, at their non-dominant wrist. In addition to wearing the accelerometer, participants will be asked to fill in a daily succinct diary with: (1) bed times, nap times; (2) non-wear times during the day; and (3) specification of most seated activity. These data will be used to complete and to explain gaps in the data set later on in the software programme. The following PA outcomes will be extracted from the ActiGraph data: average time spent per day in sedentary behaviour, light PA and moderate to vigorous PA.
Change in Physical activity & Sedentary behaviour (follow up 2) - objective: accelerometery 2 | 1 year after follow up 1; 2 years after baseline
  A second accelerometer will be placed on the right thigh, namely the activPAL (PAL Technologies Ltd, Glasgow, UK). This device measures postures due to its static acceleration and inclination features. It can quantify postural allocation - which is not possible with the ActiGraph - and is completely waterproof. The following additional PA outcomes will be extracted: time spent sitting/lying, standing, and walking.
Physical activity & Sedentary behaviour (baseline) - subjective: International Physical Activity Questionnaire - Short Form (IPAQSF) | baseline
  The IPAQ-SF is a 7-question measure that assesses frequency and duration of vigorous PA, moderate PA, walking during the past 7 days, as well as time spent sitting.
Change in Physical activity & Sedentary behaviour (follow up 1) - subjective: International Physical Activity Questionnaire - Short Form (IPAQSF) | 1 year after baseline
  The IPAQ-SF is a 7-question measure that assesses frequency and duration of vigorous PA, moderate PA, walking during the past 7 days, as well as time spent sitting.
Change in Physical activity & Sedentary behaviour (follow up 2) - subjective: International Physical Activity Questionnaire - Short Form (IPAQSF) | 1 year after follow up 1; 2 years after baseline
  The IPAQ-SF is a 7-question measure that assesses frequency and duration of vigorous PA, moderate PA, walking during the past 7 days, as well as time spent sitting.
Physical activity (baseline) - subjective: muscle strengthening activity questionnaire | baseline
  Translated version of Muscle-strengthening exercise: Assessing participation and influences - J. Shakespear-Druery, dr. J. Bennie, dr. Katrien De Cocker & prof. S. Biddle to assess frequency, intensity and duration.
Change in Physical activity (follow up 1) - subjective: muscle strengthening activity questionnaire | 1 year after baseline
  Translated version of Muscle-strengthening exercise: Assessing participation and influences - J. Shakespear-Druery, dr. J. Bennie, dr. Katrien De Cocker & prof. S. Biddle to assess frequency, intensity and duration.
Change in Physical activity (follow up 2) - subjective: muscle strengthening activity questionnaire | 1 year after follow up 1; 2 years after baseline
  Translated version of Muscle-strengthening exercise: Assessing participation and influences - J. Shakespear-Druery, dr. J. Bennie, dr. Katrien De Cocker & prof. S. Biddle to assess frequency, intensity and duration.

SECONDARY OUTCOMES:
Wellbeing (baseline) - Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) | baseline
  The 14-item scale WEMWBS has 5 response categories, summed to provide a single score
Wellbeing (follow up 1) - Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) | 1 year after baseline
  The 14-item scale WEMWBS has 5 response categories, summed to provide a single score
Wellbeing (follow up 2) - Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) | 1 year after follow up 1; 2 years after baseline
  The 14-item scale WEMWBS has 5 response categories, summed to provide a single score
Global health (baseline) - PROMIS Global health | baseline
  10-item questionnaire on health
Global health (baseline) - PROMIS Global health | 1 year after baseline
  10-item questionnaire on health
Global health (follow up 2) - PROMIS Global health | 1 year after follow up 1; 2 years after baseline
  10-item questionnaire on health
Depression (baseline) - The Geriatric Depression Scale (GDS-15) | baseline
  15-item questionnaire on depressive symptoms
Depression (follow up 1) - The Geriatric Depression Scale (GDS-15) | 1 year after baseline
  15-item questionnaire on depressive symptoms
Depression (follow up 2) - The Geriatric Depression Scale (GDS-15) | 1 year after follow up 1; 2 years after baseline
  15-item questionnaire on depressive symptoms
Loneliness (baseline) - de Jong Gierveld loneliness scale (DJG loneliness) | baseline
  The 11-item de Jong Gierveld loneliness scale is a multi-dimensional measure of loneliness and contains five positively worded and six negatively worded items. The items fall into four subscales; feelings of severe loneliness, feelings connected with specific problem situations, missing companionship, feelings of belongingness.
Loneliness (follow up 1) - de Jong Gierveld loneliness scale (DJG loneliness) | 1 year after baseline
  The 11-item de Jong Gierveld loneliness scale is a multi-dimensional measure of loneliness and contains five positively worded and six negatively worded items. The items fall into four subscales; feelings of severe loneliness, feelings connected with specific problem situations, missing companionship, feelings of belongingness.
Loneliness (follow up 2) - de Jong Gierveld loneliness scale (DJG loneliness) | 1 year after follow up 1; 2 years after baseline
  The 11-item de Jong Gierveld loneliness scale is a multi-dimensional measure of loneliness and contains five positively worded and six negatively worded items. The items fall into four subscales; feelings of severe loneliness, feelings connected with specific problem situations, missing companionship, feelings of belongingness.
Social network (baseline) - Lubben Social Network Scale (LSN-6) | baseline
  LSNS-6 provides quantitative information on their family and friendship ties, and identifies persons at increased risk for social isolation
Social network (follow up 1) - Lubben Social Network Scale (LSN-6) | 1 year after baseline
  LSNS-6 provides quantitative information on their family and friendship ties, and identifies persons at increased risk for social isolation
Social network (follow up 2) - Lubben Social Network Scale (LSN-6) | 1 year after follow up 1; 2 years after baseline
  LSNS-6 provides quantitative information on their family and friendship ties, and identifies persons at increased risk for social isolation
Expectations Regarding Aging (baseline) - 12-Item Expectations Regarding Aging survey | baseline
  12-Item Expectations Regarding Aging
Expectations Regarding Aging (follow-up 1) - 12-Item Expectations Regarding Aging survey | 1 year after baseline
  12-Item Expectations Regarding Aging
Expectations Regarding Aging (follow-up 2) - 12-Item Expectations Regarding Aging survey | 1 year after follow up 1; 2 years after baseline
  12-Item Expectations Regarding Aging

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All anonymised textual and numerical data will be available after the end of the project in an Open Access repository or upon request by mail.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Upon publication of the research results
Access Criteria: Researchers with a track record in the field of healthy ageing or physical activity and health and proven experience in the analysis of variables as collected in the study will be able to access the data.
  Data from the project that can be shared will be made available under a Creative Commons attribution license (CC-BY-NC-SA 4.0) so that users have to give credit to the original data creators.